CLINICAL TRIAL: NCT07227168
Title: A Phase 1 Open-Label Study to Evaluate Safety, Pharmacokinetics, and Preliminary Anti-Tumor Activity of STRO-004 in Adults With Refractory/Recurrent Metastatic Solid Tumors
Brief Title: A Study of STRO-004 in Adults With Refractory/Recurrent Metastatic Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sutro Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STRO-004-ST1
Record Dates: First submitted 2025-11-07; First posted 2025-11-12 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Head and Neck Squamous Cell Carcinoma HNSCC; Non-Small Cell Lung Cancer NSCLC; Esophageal Cancer; Gastric Cancer; Colorectal Cancer; Pancreatic Ductal Adenocarcinoma (PDAC); Cervical Cancer; Endometrial Cancer; Urothelial Cancer
Keywords: Tissue Factor (TF); STRO-004; Antibody Drug Conjugate; ADC
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Colorectal Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1A STRO-004 Monotherapy (Experimental)
  Interventions: Drug: STRO-004
- Part 1B STRO-004 Monotherapy (Experimental)
  Interventions: Drug: STRO-004
- Part 1C STRO-004 in Combination with Pembrolizumab (Experimental)
  Interventions: Drug: STRO-004; Drug: Pembrolizumab

INTERVENTIONS:
Drug: STRO-004 — IV Infusion
Drug: Pembrolizumab — IV Infusion
  Arms: Part 1C STRO-004 in Combination with Pembrolizumab

SUMMARY:
This is a study to evaluate the safety and preliminary anti-tumor activity of STRO-004 in adults with metastatic cancer. This study includes 3 parts:

* Part 1A is a dose escalation study of STRO-004 monotherapy in selected tumor types known to commonly express Tissue Factor (TF).
* Part 1B is a cohort expansion in 1 or more types of cancer to further evaluate a STRO-004 monotherapy dose, determine the best dose for use in later phases, and examine anti-tumor activity.
* Part 1C is a dose escalation of STRO-004 combined with pembrolizumab to determine tolerability and preliminary anti-tumor activity of both drugs used together.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented metastatic or locally advanced solid tumors including: Head and Neck Squamous Cell Carcinoma, Non-small Cell Lung Cancer, Esophageal/Gastric Cancer, Colorectal Cancer, Pancreatic Ductal Adenocarcinoma, Cervical Cancer, Endometrial Cancer, and Urothelial Carcinoma
* Age 18 years or older
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1
* Received all appropriate systemic therapies that are locally available for which they are eligible. For Parts 1A and 1C, there is no limit on the number of prior therapies. For Part 1B only, up to 3 prior therapies are allowed, except for NSCLC participants with genomic alterations, who may have up to 4 prior therapies
* Availability of tumor tissue
* Measurable disease per RECIST 1.1
* Adequate organ function
* Participants receiving anticoagulants must be on a stable dose

Exclusion Criteria:

* Eye disorders
* Untreated brain metastases
* Pre-existing clinically significant ocular disorders, active interstitial lung disease, clinically significant cardiac or cerebrovascular disease, or other significant concurrent, uncontrolled medical condition
* Previous solid organ or bone marrow transplantation
* Concurrent participation in another therapeutic treatment trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Part 1A: Number of participants with Dose-limiting Toxicities (DLTs) | Up to Day 21
Part 1A, 1B: Percentage of participants with Treatment-Emergent Adverse Events (TEAEs), with severity determined according to the Common Terminology Criteria for Adverse Events (CTCAE) v5.0 grading scale | Up to 12 Months
Part 1A, 1B, 1C: Percentage of participants with clinical laboratory abnormalities, with severity determined according to the CTCAE v5.0 grading scale | Up to 12 months
Part 1B: Objective Response Rate (ORR) | Up to 12 months
  Best response of Complete Response (CR) or Partial Response (PR) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST V1.1)
Part 1B: Disease control rate (DCR) | Up to 12 months
  The proportion of participants with best response of CR, PR or Stable Disease (SD) per RECIST V1.1
Part 1B: Duration of Response (DOR) | Up to 12 months
  Time from first occurrence of objective response to the time of Progressive Disease (PD) according to RECIST v1.1 or death from any cause, whichever comes first
Part 1B: Progression-Free Survival (PFS) | Up to 12 months
  Time from first dose to the first occurrence of PD according to RECIST v1.1 or death from any cause, whichever comes first
Part 1B: 12-month survival rate | 12 months
  Percentage of participants alive 12 months after first dose of study treatment
Part 1C: Percentage of participants with TEAEs, with severity determined according to the CTCAE v5.0 grading scale | Up to 12 months

SECONDARY OUTCOMES:
Part 1A, 1B, 1C: Plasma concentrations of STRO-004 and its metabolites at specified timepoints | Up to 12 months
Part 1A, 1B, 1C: Immunogenicity | Up to 12 months
  As measured by circulating antidrug antibody (ADA) over time
Part 1A: Objective Response Rate (ORR) | Best response of CR or PR per RECIST V1.1
  Up to 12 months
Part 1A, 1C: Disease Control Rate (DCR) | Up to 12 months
  Proportion of participants with best response of CR, PR or SD per RECIST V1.1
Part 1A, 1C: Duration of Response (DOR) | Up to 12 months
  Time from first occurrence of objective response to the time of PD according to RECIST v1.1 or death from any cause, whichever comes first
Part 1A,1C: Progression-Free Survival (PFS) | Up to 12 months
  Time from first dose to the first occurrence of PD according to RECIST v1.1 or death from any cause, whichever comes first
Part 1A,1C: 12-month survival rate | 12 months
  Proportion of participants alive 12 months after the date of first dose of study treatment

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - SCRI Denver, Denver, Colorado
  - SCRI FCS Sarasota, Sarasota, Florida
  - Mass General Cancer Center, Boston, Massachusetts
  - NEXT Austin, Austin, Texas
  - NEXT San Antonio, San Antonio, Texas
  - NEXT Virginia, Fairfax, Virginia